CLINICAL TRIAL: NCT04558541
Title: A Developmental Framework For Linking Phonological And Morpho-syntactic Sequential Pattern Rules In Developmental Language Disorder: Production
Brief Title: A Developmental Framework For Linking Phonological And Morpho-syntactic Sequential Pattern Rules In DLD: Production
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Lisa Goffman, Senior Scientist and Endowed Chair, Father Flanagan's Boys' Home
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-78
Record Dates: First submitted 2020-08-22; First posted 2020-09-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Developmental Language Disorder; Speech Sound Disorder; Specific Language Impairment
MeSH Terms: conditions — Language Development Disorders; Speech Sound Disorder; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: For children, assessments will determine group assignment. Participants will be randomly assigned to a condition, reflecting each of the 3 phonological patterns (Single Feature, OR, Family Resemblance). Randomization will occur within groups and will be generated a priori.
  Children will participate in testing and an experimental session, which includes exposure to the rule followed by a generalization test. A sub-group will participate in the Referential Study.
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers will not be told which condition they are participating in. Investigators will know because of familiarity with the stimuli.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensitivity to phonological rules: Children (Experimental): Arm 1: Single Feature Pattern; Arm 2: OR/Disjunction Pattern; Arm 3: Family Resemblance/Prototype Pattern
  Interventions: Other: Sensitivity to phonological rules
- Sensitivity to semantic category cues: Children (Experimental): Arm 1.Referential cue during OR learning.
  Interventions: Other: Sensitivity to semantic category cues.

INTERVENTIONS:
Other: Sensitivity to phonological rules — Assess whether children with developmental language disorder (DLD) are sensitive to different phonological patterns that are predicted to align with development of morphosyntax or the lexicon; children with speech sound disorder (SSD) are not predicted to be sensitive to the same phonological patterns.
  Arms: Sensitivity to phonological rules: Children
Other: Sensitivity to semantic category cues. — Assess whether all children, including those with DLD, show improved learning of OR rules when a semantic category cue is used.
  Arms: Sensitivity to semantic category cues: Children

SUMMARY:
The broad aim of this clinical study is to assess the hypothesis that morphological and phonological deficits are linked by a broader deficit in sequential pattern learning. This hypothesis applies to learning in general, but is especially critical as an avenue for developing earlier assessments and more powerful interventions for children with developmental language disorder (DLD; also known as specific language impairment). Other populations, such as at-risk toddlers, may also benefit from this new approach.

DETAILED DESCRIPTION:
The developmental approach taken here combines what is already known about morpho-syntactic deficits in DLD with recent developments in the fields of linguistics and language acquisition. First, it is possible to divide phonological and morphological patterns into three pattern types (Single Feature, OR/Disjunction, Family Resemblance/Prototype), with these types having a long history of study in visual pattern learning. Importantly, children with DLD appear to have maximum difficulty with morpho-syntactic patterns of the OR type (e.g., regular past tense; add a "t" if the final consonant is voiceless OR a "d" if the final consonant is voiced). In contrast, studies using artificial grammars show that infants who are typically developing are highly adept at learning Single Feature and OR pattern types; Family Resemblance patterns may be weaker. Family resemblance patterns relate to similarity, and may be more closely tied to the lexicon than to grammar (e.g., beagles and terriers are similar and they are both dogs; the words "goat" and "boat" are similar). Typical adults are adept at Single Feature and Family Resemblance patterns, but appear to be, at least superficially, more like children with DLD in their performance on the OR pattern.

With these developmental findings as a starting point, the proposed research links phonological and morphological sequence learning in children with developmental language disorder (DLD). In the studies focused on children, the investigators ask if 4- to 6-year-olds who are typically developing as well as those with DLD (both with and without co-occurring speech sound deficits) and speech sound disorder (SSD; without co-occurring morpho-syntactic deficits) are sensitive to input examples that fit one of these three patterns. The hypothesis is that, consistent with their long-documented morpho-syntactic deficit, children with DLD will have particular difficulty with the OR pattern. Consistent with their intact morpho-syntactic skills, children with SSD should show no deficits in the OR pattern, revealing a link between OR pattern learning, phonology, and morpho-syntax. The endpoint measure is that children with DLD (both with and without an accompanying SSD) do not show sensitivity to the OR pattern, as measured by sound pattern (e.g., phonetic accuracy, syllable sequence stability) and motor learning (e.g., articulatory and acoustic variability) measures.

This hypothesis is assessed by indexing the learning trajectory across the training period and during generalization to new nonwords that are consistent or inconsistent with the training pattern. In the generalization phase, children are asked to name new novel words that are either consistent (i.e., that fit the training rule) or inconsistent (i.e., that do not fit the training rule) nonwords. It is predicted that children with TD and SSD, who are still in a period of language learning plasticity (they can still learn the sound patterns and grammar of a second language) will be sensitive to all three patterns. However, children with DLD (both with and without accompanying SSD) are predicted to show sensitivity to the family resemblance and single feature patterns, but not to the critical OR pattern-the one associated with sound pattern and grammatical learning, This would reveal an important connection between sound pattern and grammatical learning, which could lead to earlier diagnosis (phonological patterns emerge earlier than grammar) and to more general intervention practices that focus on sequential pattern learning rather than specific language goals may be efficacious.

A second aim explores whether the inclusion of a semantic subcategory cue facilitates learning the OR pattern. The hypothesis is that children with DLD (as well as typical adults) who initially are predicted to have the most difficulty with the OR pattern, will show increases in sensitivity following the addition of a semantic category cue (e.g., animals for the voiced consonant rule OR tools for the voiceless consonant rule). This result would be especially important for learners with DLD, as it may provide a pathway for intervention of a core learning deficit.

Critically, these studies are developmental in nature. In the adult component of this research (conducted under a separate clinical trial, Gerken, University of Arizona), the investigators ask if adults are sensitive to input examples that fit one of these three patterns. The hypothesis, based on previous findings from the Gerken lab, is that adults, like children with DLD, do not show sensitivity to the OR pattern. However, adults are sensitive to single feature and Family Resemblance patterns. Adults still learn words readily and are sensitive to family resemblance prototype relationships. For adults, perceptual measures index sensitivity. Similar to the children with typical development, DLD and SSD, the investigators explore whether the inclusion of a semantic subcategory cue facilitates learning the OR pattern in adults. The hypothesis is that all learners, including adults, will show increases in sensitivity following the addition of a semantic category cue (e.g., animals for voiced rule OR tools for voiceless rule). The findings from adults contribute to a dynamic developmental framework. Because of the dramatic developmental changes in sensitivity to phonological sound patterns and the presumed linkage of such patterns to morpho-syntax, the data from adults are essential in identifying the underlying mechanism(s) of DLD and to suggesting possible intervention strategies, such as employing semantic cues to the OR pattern and strengthening lexical organization.

From previous work, it is known that infants are sensitive to the OR rule. In the studies focused on toddlers (also in a separate clinical trial conducted by Gerken at the University of Arizona), the investigators ask if dependence on the associatively organized lexicon can account for the infant-to-adult developmental changes observed for the OR pattern (which is not associatively organized) and thereby explores the possibility that children with DLD rely on their lexicons to compensate for their sequential pattern learning deficit. The hypothesis is that 20-month-old children, who are just entering a period of rapid vocabulary learning, will show increased sensitivity (based on looking time to words that are consistent vs. inconsistent within the training set) in the family resemblance condition when a visual referent (i.e., semantic cue) is added, but decreased sensitivity in the OR condition when a visual referent is added. These results will also be related to vocabulary size as reported on the MacArthur-Bates Communicative Development Inventory, with the prediction that robust patterns are smaller for children who received referents or who have smaller vocabularies for the OR pattern and greater for children who received referents or who have larger vocabularies for the family resemblance pattern. The results from toddlers, who are just entering a period of rapid vocabulary learning, provide an essential framework for understanding how different types of phonological patterns apply to lexical and morpho-syntactic learning.

The results of the proposed studies provide a critical developmental framework for identifying the underlying mechanism(s) of DLD. These findings will also lead to the development of intervention strategies, such as strengthening lexical organization, to support problematic aspects of sequential pattern learning.

ELIGIBILITY:
Inclusion Criteria:

Because clinical precision is required, 4- to 8-year-olds will complete a large test battery.

* All children (TD, DLD, DLD + SSD, SSD) will score above 75 on the Nonverbal Scale of the Kaufman Assessment Battery for Children (KABC-II), which is above the Diagnostic and Statistical Manual cut-off for intellectual disability, even considering the standard error of measurement.
* Hearing will be within normal limits
* Oral structures will be within normal limits (Robbins & Klee, 1987).
* The Childhood Autism Rating Scale (Schopler et al., 2010) and parent report, will be used to rule out autism.

Children with DLD will meet standard criteria.

* Children with DLD will score below the cutoff of 87 on the Structured Photographic Expressive Language Test-P2 (SPELT-P2; Dawson et al., 2005) that has demonstrated high diagnostic accuracy for DLD.
* Children with DLD will perform below 80% in their spontaneous production of finite verb morphemes.
* Performance on a nonword repetition task will also support DLD status. Scores below 70% for total phonemes correct across all nonword lengths are greater than 1 SD below the mean for typical children.
* Speech production skills will be measured via the Goldman-Fristoe Test of Articulation-3 (GFTA-3; Goldman & Fristoe, 2015) and the inconsistency subtest of the Diagnostic Evaluation of Articulation and Phonology (DEAP, Dodd, et al., 2006). Many 4- to 6-year-old children with DLD are expected to perform below expected levels on the GFTA-3; for this study half of the children with DLD will show performance below expected levels and half above a standard score of 85. Children with SSD will show impaired performance on the GFTA-3, but typical performance on grammatically weighted language measures (SPELT-P2 and finite verb morphemes). The DEAP serves as a standardized measure of segmental inconsistency and will provide a post hoc analysis that may be related to sequence pattern variability.

Performance on the following measures will serve as covariates and will not be exclusionary for DLD or SSD:

* Peabody Picture Vocabulary Test, 4th ed (Dunn & Dunn, 1997)
* Expressive Vocabulary Test, 2nd ed (Williams, 1997)
* Verbal and nonverbal memory span.
* Because of the emphasis on English phonological and morpho-syntactic patterns, all participants will be monolingual English learners or report dominant exposure to English from infancy. Exposure to other languages will be documented.

Exclusion Criteria for all participants:

* Hearing impairment
* Intellectual impairment
* Autism
* Significant motor impairment.

Typical participants will be excluded if they show:

-Histories of developmental, speech, language, or hearing disorders.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2022-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcription Accuracy Measures of Children's Sensitivity to OR/disjunction, Family resemblance/prototype and/or Single feature rules | 30 minutes
  Learning shown via changes in transcription accuracy
Transcription Variability Measures of Children's Sensitivity to OR/disjunction, Family resemblance/prototype and/or Single feature rules | 30 minutes
  Learning shown via changes in transcription based syllable co-occurrence variability
Articulatory Variability Measures of Children's Sensitivity to OR/disjunction, Family resemblance/prototype and/or Single feature rules | 30 minutes
  Learning shown via changes in articulatory variability (articulatory spatiotemporal variability)
Acoustic Measures of Children's Sensitivity to OR/disjunction, Family resemblance/prototype and/or Single feature rules | 30 minutes
  Learning shown via changes in acoustic variability (Acoustic spatiotemporal variability)
Transcription Accuracy Measures of Children's Sensitivity to OR/disjunction with the inclusion of a semantic category cue. | 30 minutes
  Learning shown via changes in transcription accuracy
Transcription Variability Measures of Children's Sensitivity to OR/disjunction with the inclusion of a semantic category cue. | 30 minutes
  Learning shown via changes in transcription based syllable co-occurrence variability
Articulatory Variability Measures of Children's Sensitivity to OR/disjunction with the inclusion of a semantic category cue. | 30 minutes
  Learning shown via changes in articulatory variability (articulatory spatiotemporal variability)
Acoustic Variability Measures of Children's Sensitivity to OR/disjunction with the inclusion of a semantic category cue. | 30 minutes
  Learning shown via changes in acoustic variability (acoustic spatiotemporal variability)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Boys Town National Research Hospital, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No